CLINICAL TRIAL: NCT00559884
Title: An Open-label, Randomized, Single Dose, Crossover Study to Assess the Pharmacokinetics, Pharmacodynamics, Safety, and Tolerability of Modified Release Formulations of GSK189075 in Healthy Volunteers
Brief Title: A Study to Compare the Safety and Drug Levels in Blood When Using Various Forms of GSK189075 Given to Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: KGW111057
Record Dates: First submitted 2007-11-14; First posted 2007-11-16 (Estimated); Last update posted 2012-06-04 (Estimated); Status verified 2011-02

CONDITIONS: Type 2 Diabetes Mellitus; Diabetes Mellitus, Type 2
Keywords: pharmacokinetics,; healthy male and females,; pharmacodynamics
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: GSK189075 (Modified and immediate release formulations)

SUMMARY:
The purpose of this research study is to look at concentrations of GSK189075 in blood when different long and short acting forms of the drug are taken by mouth. The results will help to decide whether a long-acting form of GSK189075 can be made. The effects of the drug on the body and safety will also be studied.

ELIGIBILITY:
Inclusion Criteria:

* Are a healthy, non-smoking adult, 18 to 55 years old.
* Are not overly thin or overly heavy for your height.
* Are a female who is unable to have children, or is willing to use birth control throughout the study.
* Are willing and able to follow all study-related instructions provided by the site staff. - Are willing to provide signed consent.

Exclusion Criteria:

* Are a pregnant or a nursing female.
* Have a past or current disease such as heart, liver, kidney, blood, brain, or other disease.
* Have had certain infections within 4 weeks before the expected the first dose of study drug.
* Have HIV or hepatitis, or have alcohol in your system at the screening visit.
* Have a history of alcohol abuse.
* Have been in another research study in the last month or have taken certain medications in the 2 weeks before study drug would be taken.
* Have laboratory tests that are outside the normal range.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2007-11

PRIMARY OUTCOMES:
Blood samples: | collected over 24-hour period after each different form of GSK189075 given to measure amount of drug in blood
Urine: | collected over 24-hour period after dosing with each form to measure amount of urine produced & amount of sugar in urine

SECONDARY OUTCOMES:
Adverse events: | all visits after Day -1
blood pressure & heart rate: | screening,Day -1 - Day 1,follow-up visit
ECGs: | screening,pre-dose, Day 1
lab tests: | screening, Day -1 - Day 1,follow-up

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Columbus, Ohio, United States